CLINICAL TRIAL: NCT06857435
Title: Autologous Point-of-Care Adipose Therapy for Reconstruction and Regeneration of Traumatized Skin: Delayed Injury/Scar
Brief Title: Autologous Point-of-Care Adipose Therapy: Delayed Injury/Scar
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Armed Forces Institute of Regenerative Medicine (U.S. Federal Agency)
Responsible Party: Principal Investigator, Francesco Egro, Director of Burn Reconstruction, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY24080150 - Delayed Injury
Record Dates: First submitted 2025-02-04; First posted 2025-03-04 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-11

CONDITIONS: Burns; Contracture Scar; Surgical Injury
Keywords: burns; scar contracture
MeSH Terms: conditions — Burns; Intraoperative Complications | interventions — Plastic Surgery Procedures

STUDY DESIGN:
Intervention Model Description: Autologous Layered Composite Grafting consists of the layered strategy of simultaneous fat and skin grafting. Fat is harvested by minimally invasive liposuction and applied directly to the wound base without any chemical or biologic processing. Skin is harvested as per standard of care and applied either to the wound bed directly as per controls or to the layer of adipose tissue.
  Investigators will compare delayed reconstruction of scar contracture across two treatment arms (40 subjects).
  * Group 1: Full thickness skin graft (FTSG) Reconstruction;
  * Group 2: Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Grafting).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Full Thickness Skin Graft (FTSG) Reconstruction (Active Comparator): In this Arm, the investigators will assess FTSGs for reconstruction of defects after burn scar revision of the face, neck, or extremities. Participants will receive any release and/or preparation of the scar/wound bed as would be standard of care and will then receive reconstruction with a FTSG.
  Interventions: Procedure: Full Thickness Skin Graft (FTSG)
- Delayed Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Graft) (Experimental): In this Arm, the investigators will assess Autologous Layered Composite Grafting for reconstruction of defects after burn scar revision of the face, neck, or extremities. Participants will receive any release and/or preparation of the scar/wound bed as would be standard of care and will then receive reconstruction with a Autologous Layered Composite Graft.
  Interventions: Procedure: Base of wound fat graft with Split Thickness Skin Graft (STSG) Reconstruction (Autologous Layered Composite Grafting).

INTERVENTIONS:
Procedure: Full Thickness Skin Graft (FTSG) — Full thickness skin in FTSGs are harvested by different means by surgeon preference and standard of care. Typically an area of skin with matching color and texture to the site which needs reconstruction is identified from a hidden and/or non-cosmetic area and collected via excision. After excision the donor site is closed and the graft is thinned by using a scalpel or scissors to remove excess fat or other soft tissues from the deep surface before being placed in the donor site.
  Arms: Delayed Full Thickness Skin Graft (FTSG) Reconstruction
Procedure: Base of wound fat graft with Split Thickness Skin Graft (STSG) Reconstruction (Autologous Layered Composite Grafting). — Autologous Layered Composite Grafting consists of the layered strategy of simultaneous fat and skin grafting. Fat is harvested by minimally invasive liposuction and applied directly to the wound base without any chemical or biologic processing. Skin is harvested as a split thickness skin graft by dermatome and applied over the layer of adipose tissue.
  Arms: Delayed Base of wound fat graft with STSG Reconstruction (Autologous Layered Composite Graft)

SUMMARY:
The goal of this study is to explore if an adipose-based therapeutic strategy can treat contracted scars secondary to soft-tissue burn wounds in injured individuals, especially those with severe burns or soft-tissue loss. The main question it aims to answer are:

- Can autologous layered composite grafting demonstrate non-inferiority compared to full-thickness skin grafting for delayed reconstruction of post-burn or trauma scar contracture?

Researchers will compare the single-stage autologous layered composite grafting method to traditional methods to see if it improves healing outcomes, minimizes scarring, and reduces infection risk.

Participants will:

* Receive fat grafting at time of scar revision.
* Undergo simultaneous split-thickness skin grafting for full soft-tissue reconstruction.

DETAILED DESCRIPTION:
Soft-tissue injuries from blasts, burns, or multiple traumas can cause severe damage, leading to loss of function, lower quality of life, long recovery times, and inability to work. When these injuries involve deep burns or full-thickness tissue loss in areas that move a lot, they are especially difficult to treat due to the risk of scarring, stiffness, and tissue sticking together. There is a need for a reliable, single-stage treatment that can provide soft, flexible tissue reconstruction with minimal risk, cost, and, complexity. To address this issue, the investigators propose a fat-based approach to reconstruction. Fat tissue is easily available from the patient's own body and carries many benefits in reconstructive surgery. Our team has shown that using a layer of fat immediately in treatment creates a soft, vascular layer that reduces scarring, improves tissue volume, and supports a one-stage, multi-layer reconstruction without the need for complex surgery or causing harm to the donor area. The purpose of this study is to compare this reconstructive approach under the following conditions:

• Demonstrate non-inferiority of autologous layered composite grafting to full-thickness skin grafting for delayed reconstruction of post-burn/trauma scar contracture.

Evaluators including dedicated observers will be blinded to treatment group/strategy.

ELIGIBILITY:
Inclusion Criteria:

* The proposed study will include adult patients 18 years of age or older,
* male or female,
* civilian, military, active duty or retired veterans
* presenting for scar contracture release and reconstruction at any level.
* Additional inclusion criteria includes willingness to be randomized to receive a fat graft.

Exclusion Criteria:

* Age < 18 years of age,
* active infection,
* medical co-morbidities or anatomic configuration deemed by the physician to be a concern for safety,
* unwilling or unable to comply with study procedures,
* radiation to the site of interest,
* prisoners and/or vulnerable populations.
* In addition, candidates that are pregnant or plan to become pregnant in the next year, will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-01-31 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
Change in scar contracture, as measured by change in scar surface area size | From surgery to 9-month clinical endpoint.
  Contracture as measured by change in surface area of reconstruction between time of surgery and 9-month clinical endpoint/maturation of reconstruction. These data will be derived by serial photography.

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability). | From surgery to 9-month clinical endpoint.
  Incidence of adverse events will be reported for all study participants.
Total score on the Patient and Observer Scar Assessment Scale (POSAS): Pigmentation, Pliability, Vascularity, Thickness, Relief, and Surface Area, collected at the 9 month follow up visit. Remove | From surgery to 9-month clinical endpoint.
  POSAS measures subjective assessment on a 1-10 scale from normal skin to worst scar imaginable across 6 metrics (surface area, vascularity, pigmentation, thickness, pliability and relief). The lowest sum score, reflecting normal skin, is 6 and the highest score, reflecting the worst imaginable scar, is 60.
Number of Operative Encounters | From surgery to 9-month clinical endpoint.
  The investigators will additionally assess early outcome metrics including number of operative encounters.
Percent Graft Take | From surgery to 9-month clinical endpoint.
  The investigators will additionally assess early outcome metrics including percent graft take (% of surface area).
Time to Final Healing/Graft Take | From surgery to 9-month clinical endpoint.
  The investigators will additionally assess early outcome metrics including, time to final healing/graft take in days.
Tissue Thickness | From surgery to 9-month clinical endpoint.
  The investigators will measure tissue thickness as determined by ultrasound.
Pliability (Tensiometry/Cutometry) | From surgery to 9-month clinical endpoint.
  The investigators will utilize a noninvasive cutometer/tensiometer to determine tissue pliability.
Tissue Adhesion/Mobility | From surgery to 9-month clinical endpoint.
  The investigators will measure tissue mobility/resistance to adhesion under non-invasive tissue stretch.

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Egro, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Mercy Hospital, Pittsburgh, Pennsylvania
  - Presbyterian Hospital, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piccolo NS, Piccolo MS, Piccolo MT. Fat grafting for treatment of burns, burn scars, and other difficult wounds. Clin Plast Surg. 2015 Apr;42(2):263-83. doi: 10.1016/j.cps.2014.12.009. Epub 2015 Feb 21. PMID 25827568
- [Background] Simonacci F, Bertozzi N, Grieco MP, Grignaffini E, Raposio E. Procedure, applications, and outcomes of autologous fat grafting. Ann Med Surg (Lond). 2017 Jun 27;20:49-60. doi: 10.1016/j.amsu.2017.06.059. eCollection 2017 Aug. PMID 28702187
- [Background] Evans BGA, Gronet EM, Saint-Cyr MH. How Fat Grafting Works. Plast Reconstr Surg Glob Open. 2020 Jul 14;8(7):e2705. doi: 10.1097/GOX.0000000000002705. eCollection 2020 Jul. PMID 32802628
- [Background] Woodruff SI, Galarneau MR, McCabe CT, Sack DI, Clouser MC. Health-related quality of life among US military personnel injured in combat: findings from the Wounded Warrior Recovery Project. Qual Life Res. 2018 May;27(5):1393-1402. doi: 10.1007/s11136-018-1806-7. Epub 2018 Feb 15. PMID 29450855
- [Background] Mokos ZB, Jovic A, Grgurevic L, Dumic-Cule I, Kostovic K, Ceovic R, Marinovic B. Current Therapeutic Approach to Hypertrophic Scars. Front Med (Lausanne). 2017 Jun 20;4:83. doi: 10.3389/fmed.2017.00083. eCollection 2017. PMID 28676850
- [Background] Finnerty CC, Jeschke MG, Branski LK, Barret JP, Dziewulski P, Herndon DN. Hypertrophic scarring: the greatest unmet challenge after burn injury. Lancet. 2016 Oct 1;388(10052):1427-1436. doi: 10.1016/S0140-6736(16)31406-4. PMID 27707499
- [Background] Marshall CD, Hu MS, Leavitt T, Barnes LA, Lorenz HP, Longaker MT. Cutaneous Scarring: Basic Science, Current Treatments, and Future Directions. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):29-45. doi: 10.1089/wound.2016.0696. PMID 29392092
- [Background] Wolf JM, Athwal GS, Shin AY, Dennison DG. Acute trauma to the upper extremity: what to do and when to do it. Instr Course Lect. 2010;59:525-38. PMID 20415403
- [Background] Harrison BL, Lakhiani C, Lee MR, Saint-Cyr M. Timing of traumatic upper extremity free flap reconstruction: a systematic review and progress report. Plast Reconstr Surg. 2013 Sep;132(3):591-596. doi: 10.1097/PRS.0b013e31829ad012. PMID 23676968
- [Background] Le TD, Gurney JM, Nnamani NS, Gross KR, Chung KK, Stockinger ZT, Nessen SC, Pusateri AE, Akers KS. A 12-Year Analysis of Nonbattle Injury Among US Service Members Deployed to Iraq and Afghanistan. JAMA Surg. 2018 Sep 1;153(9):800-807. doi: 10.1001/jamasurg.2018.1166. PMID 29847675
- [Background] D'Souza EW, MacGregor AJ, Dougherty AL, Olson AS, Champion HR, Galarneau MR. Combat injury profiles among U.S. military personnel who survived serious wounds in Iraq and Afghanistan: A latent class analysis. PLoS One. 2022 Apr 6;17(4):e0266588. doi: 10.1371/journal.pone.0266588. eCollection 2022. PMID 35385552